CLINICAL TRIAL: NCT01113307
Title: A Multi-Center Post- Marketing Study to Define Procedures for the Use of CureXcellTM in a Community Setting for the Treatment of Wounds
Brief Title: The Use of CureXcellTM in a Community Setting for the Treatment of Hard to Heal Wounds
Status: Completed | Type: Observational
Sponsor: Macrocure Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: MC-103
Record Dates: First submitted 2010-04-28; First posted 2010-04-29 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Wounds
Keywords: Chronic ulcers; pressure ulcers; venous ulcers; diabetic foot ulcers; post operative ulcers; hard to heal ulcers
MeSH Terms: conditions — Wounds and Injuries; Pressure Ulcer; Varicose Ulcer; Diabetic Foot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hard to heal wounds
  Interventions: Biological: Activated allogeneic white blood cells

INTERVENTIONS:
Biological: Activated allogeneic white blood cells — The CUREXCELL™ dosage form consists of an activated cell suspension that has been isolated, activated and purified from the peripheral blood of healthy allogeneic donors, by hypo-osmotic shock, using the MacroCure custom closed bag system.The cell suspension is superficially injected throughout the wound bed ( 0.1ml per 1 cm2 of wound bed).
  Other Names: CureXcell

SUMMARY:
The primary objective of the study is to define procedures for the use of CureXcellTM in the community through Clalit Health Services. Secondary objective is to evaluate the blinding method in a subgroup of patients, which will be used in a future study named: a multinational, multi-center, randomized, double blind, placebo controlled study for the evaluation of the tolerability, safety and efficacy of CureXcell™ therapy plus adequate ulcer treatment, in diabetic patients with ulcers in the lower extremities.

Adults with chronic ulcers; pressure ulcers, venous ulcers, diabetic foot ulcers or post operative ulcer will be recruited to the study. Patients that have been recruited for the study will be treated as required for their medical condition. As required, cultures will be taken, IV or PO antibiotics will be given and debridement will be carried out. Patients will be referred to catheterization, revascularization, or amputation as required and the decision to do so will not be affected in any way by the study. CureXcellTM will be used as adjunct treatment to good ulcer care (GUC).

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 18 and 90 years of age with one ulcer that has not shown signs of normal healing (according to physician experienced in wound therapy) for more than 3 weeks
2. The patient suffers from diabetic ulcer, decubitus ulcer, venous insufficiency ulcer and post operative wound.
3. In patients with suspected malnutrition albumin > 2.5 g/dL in blood tests performed within the last three weeks.
4. Patients with adequate blood perfusion: palpated distal pulses TP or DP or if not palpable, arterial pressures during rest ABI > 0.6.
5. Patients without edema over +2 (patient's edema must be controlled by medical and/or bandaging or lympha press).
6. Use of elastic bandaging in wounds due to venous insufficiency (when there is no involvement of an arterial problem).
7. Wound condition does not immediately jeopardize the extremity.
8. The patient's life is not at risk (for any reason).
9. The Patient has a life expectancy of at least one year.
10. Women of childbearing potential must be willing to use reliable methods of birth control.
11. Willing and able to sign an informed consent form and attend the follow up according to the treating staff instructions until complete wound closure.

Inclusion criteria in the 'treatment blinding guessing test':

1. A patient suffering from diabetes and a chronic ulcer in the lower extremity (ankle and below) and is CureXcell™ -naive.
2. Signing an appendix to the consent form for the 'treatment blinding guessing test'.

Exclusion Criteria:

1. More than one wound;
2. Inadequately treated recurrent pressure components in the wound. If required, ulcer will be treated with preliminary treatment for local pressure components (shoes and even cast or wheel chair for the treatment period)
3. Neoplastic ulcer
4. A patient with active malignant disease during the last five years, except for a patient suffering from adequately treated Basal Cell Carcinoma which does not present in the wound area.
5. Sepsis
6. Confirmed osteomyelitis
7. Patients suffering from significant immunosuppression.
8. INR > 3 in patients receiving anticoagulation drugs, in blood tests performed within two weeks prior to the first injection
9. A response to previous blood infusions (in case administered)
10. Patient receiving unique blood components (radiated, washed etc.)
11. Pregnant patient
12. Wounds for more than a year
13. A fistula/cavity which anatomical shape does not enable a direct injection into the wound
14. A patient participating in another clinical trial, or who participated in another clinical trial within the last 30 days.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with chronic ulcers; pressure ulcers, venous ulcers, diabetic foot ulcers or post operative ulcers.
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2010-05; Primary Completion 2011-07 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with complete wound closure | Week 24

SECONDARY OUTCOMES:
Median time to complete wound closure | End of study
Change in wound area between Baseline and Last Observation | End of study
Rate of wound infections, cellulitis, and osteomyelitis | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Ram Avrahami, MD, Principal Investigator — Clalit Health Services; David Snir, MD, Principal Investigator — Clalit Health Services; Yibgeni Sherman, MD, Principal Investigator — Clalit Health Services; David Vigoda, MD, Principal Investigator — Clalit Health Services; Dimitri Gimelreich, MD, Principal Investigator — Clalit Health Services; Asher Corcos, MD, Principal Investigator — Clalit Health Services; Laios Kazir, MD, Principal Investigator — Clalit Health Services
Locations (7):
- Israel (7):
  - Omer Clalit Clinic, Afula
  - Sold Clalit Clinic, Beersheba
  - Hamoshava Diabetic Wound Clinic, Jerusalem
  - Ramat Eshcol Wound Clinic, Jerusalem
  - Zvulun Wound Clinic, Kiryat Bialik
  - Hasharon Medical Center, Petah Tikva
  - Zamenhoff Wound Clinic, Tel Aviv